CLINICAL TRIAL: NCT05264324
Title: The Impact of Hypoxia on Patients With Precapillary Pulmonary Hypertension and Treatment of Adverse Effects
Brief Title: Maximal Exercise Capacity at 2500 m of High Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: OVERALP II D
Record Dates: First submitted 2021-10-14; First posted 2022-03-03 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: High Altitude Pulmonary Hypertension; Maximal Exercise Capacity
MeSH Terms: conditions — Pulmonary edema of mountaineers

STUDY DESIGN:
Intervention Model Description: Patients will be exposed to ambient air at 490m vs. hypoxic air at 2500m in a randomized sequence according to a cross-over design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High altitude 2500 m above sea level (high altitude) (Experimental): Maximum Exercise Capacity in high altitude
  Interventions: Procedure: Maximal Exercise Capacity
- Low altitude 470 m above sea level (low altitude) (Active Comparator): Maximum Exercise Capacity in low altitude
  Interventions: Procedure: Maximal Exercise Capacity

INTERVENTIONS:
Procedure: Maximal Exercise Capacity — Maximal Exercise Capacity in incremental ramp exercise tests.

SUMMARY:
The impact of hypoxia on maximal work rate during incremental ramp exercise within 3-6 hours after arriving at 2500m of high altitude in patients with precapillary pulmonary hypertension

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature (Appendix Informed Consent Form)
* PH class I (PAH) or IV (CTEPH) diagnosed according to guidelines: mean pulmonary artery pressure >20 mmHg, pulmonary vascular resistance ≥3 wood units, pulmonary arterial wedge pressure ≤15 mmHg during baseline measures at the diagnostic right-heart catheterization

Exclusion Criteria:

* resting partial pressure of oxygen <8 kilopascal at Zurich at 490 m low altitude
* exposure to an altitude >1000 m for ≥3 nights during the last 2 weeks before the study
* inability to follow the procedures of the study
* other clinically significant concomitant end-stage disease (e.g., renal failure, hepatic dysfunction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Maximal work rate | 30 hours
  Change in maximal work rate in Watt at 2500 vs. 490 m

SECONDARY OUTCOMES:
Heart rate | 30 hours
  Change in cardiorespiratory measurements: heart rate during a cycle incremental ramp exercise test at high altitude vs. low altitude
Ventilation | 30 hours
  Change in cardiorespiratory measurements: ventilation during a cycle incremental ramp exercise test at high altitude vs. low altitude
Oxygen uptake | 30 hours
  Change in cardiorespiratory measurements: Oxygen uptake, SpO2, blood gases during a cycle incremental ramp exercise test at high altitude vs. low altitude
Arterial blood oxygenation saturation | 30 hours
  Change in cardiorespiratory measurements: Oxygenation (SpO2) during a cycle incremental ramp exercise test at high altitude vs. low altitude
Blood gases | 30 hours
  Change in blood gases during a cycle incremental ramp exercise test at high altitude vs. low altitude
Hemodynamics | 30 hours
  Change in hemodynamics assessed by echocardiography
Borg dyspnoea and leg fatigue scale | 30 hours
  Change in post-exercise Borg dyspnoea and leg fatigue scale during a cycle incremental ramp exercise test at high altitude vs. low altitude
Visual Analogue Scale for dyspnea | 30 hours
  Change Visual Analogue Scale at high altitude vs. low altitude according to a 10cm scale from left to right, where the subject has to mark dyspnea with higher values in cm meaning worse dyspnea
Electro cardiography | 30 hours
  Prevalence of abnormal resting electro cardiography (ECG) at high altitude vs. low altitude
Electro cardiography :ST-segment changes | 30 hours
  Difference in ST-segment changes during cycle incremental ramp and constant work-rate exercise tests at high altitude vs. low altitude
Electro cardiography: ST-segment changes under oxygen | 30 hours
  7Difference in ST-segment changes during cycle exercise tests without and with oxygen at high altitude
Electro cardiography: Clinically relevant ischemia | 30 hour
  Incidence of clinically relevant ischemia (>1mm ST-segment depression) during cycle exercise tests at high altitude vs. low altitude
Electro cardiography: QT-Interval | 30 hours
  Change of corrected QT-Interval, during cycle exercise tests at high vs. low altitude
Electro cardiography: QT-Interval | 30 hours
  Change of corrected QRS duration, during cycle exercise tests at high vs. low altitude
Electro cardiography: PQ-Interval | 30 hours
  Change of corrected PQ-Interval, during cycle exercise tests at high vs. low altitude
Rate pressure product | 30 hours
  Change of corrected Rate pressure product, during cycle exercise tests at high vs. low altitude
Electro cardiography: Cardiac arrhythmia | 30 hours
  Incidence of cardiac arrhythmia during cycle exercise tests at high altitude vs. low altitude

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory Clinic, University Hospital of Zurich, Zurich, Switzerland